CLINICAL TRIAL: NCT06230159
Title: Synthetic Cooling Agents in Combustible Cigarettes: A Pilot Study
Brief Title: Evaluating the Impact of Synthetic Cooling Agents in Combustible Cigarettes on Smoking Perceptions and Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Alayna Tackett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: OSU-23208; NCI-2023-10761 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-01-04; First posted 2024-01-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Spirometry

STUDY DESIGN:
Intervention Model Description: Using a cross-over double-blinded study design, we will study the abuse liability (including sensory characteristics and appeal) of newly introduced cooling agent non-menthol cigarettes.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and data collection staff will be blinded to the order/conditions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Menthol cigarette (Active Comparator): Participants participate in an ad libitum smoking session with a menthol cigarette for this condition. Participants also participate in an ad libitum smoking session with either their usual brand cigarette or the menthol study cigarette at the end of each study visit.
  Interventions: Behavioral: Menthol Cigarette Smoking; Behavioral: Usual Brand Cigarette Smoking; Diagnostic Test: Spirometry; Other: Questionnaire Administration; Diagnostic Test: Nasal Epithelial Lining Fluid
- Non-menthol cigarette (Active Comparator): Participants participate in an ad libitum smoking session with a non-menthol control cigarette for this condition. Participants also participate in an ad libitum smoking session with either their usual brand cigarette or the non-menthol study cigarette at the end of each study visit.
  Interventions: Behavioral: Non-menthol Cigarette Smoking; Behavioral: Usual Brand Cigarette Smoking; Diagnostic Test: Spirometry; Other: Questionnaire Administration; Diagnostic Test: Nasal Epithelial Lining Fluid
- Cigarette with synthetic cooling agents (Active Comparator): Participants participate in an ad libitum smoking session with a synthetic cooling agent cigarette for this condition. Participants also participate in an ad libitum smoking session with either their usual brand cigarette or the synthetic cooling agent study cigarette at the end of each study visit.
  Interventions: Behavioral: Synthetic Cooling Agent Cigarette Smoking; Behavioral: Usual Brand Cigarette Smoking; Diagnostic Test: Spirometry; Other: Questionnaire Administration; Diagnostic Test: Nasal Epithelial Lining Fluid

INTERVENTIONS:
Behavioral: Non-menthol Cigarette Smoking — Smoke a non-menthol cigarette
  Arms: Non-menthol cigarette
Behavioral: Menthol Cigarette Smoking — Smoke a menthol cigarette
  Arms: Menthol cigarette
Behavioral: Synthetic Cooling Agent Cigarette Smoking — Smoke a synthetic cooling agent cigarette
  Arms: Cigarette with synthetic cooling agents
Behavioral: Usual Brand Cigarette Smoking — Smoke usual brand cigarette
Diagnostic Test: Spirometry — Pulmonary function test
Other: Questionnaire Administration — Survey questionnaires
Diagnostic Test: Nasal Epithelial Lining Fluid — Nasal strip inserted into the nare to collect nasal epithelial lining fluid.

SUMMARY:
This clinical trial evaluates the impact of synthetic cooling agents in combustible cigarettes on smoking perceptions and use. Menthol, a natural chemical, is a cooling agent that increases nicotine dependence among smokers. Menthol cigarettes largely contribute to the huge burden that smoking puts on public health. Approximately 43% of adult smokers smoke menthol cigarettes. Regulatory agencies have begun a ban on menthol. In response to the ban, the tobacco industry has introduced synthetic cooling agents as a flavorless replacement to provide the same cooling effects as menthol. Information gained from this trial may help researchers determine how the addition of synthetic cooling agents changes the appeal, abuse liability potential, and respiratory toxicity profile of combustible cigarettes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the content of synthetic cooling agents in newly introduced cooling agent non-menthol, menthol, and traditional non-menthol cigarettes.

II. Assess the subjective effects and abuse liability of cooling agent non-menthol cigarettes.

EXPLORATORY OBJECTIVE:

I. Examine acute changes to pulmonary health associated with cooling agent cigarette use.

OUTLINE: Participants are randomized to use 1 of 3 cigarette conditions at 3 different study visits.

Participants participate in ad libitum smoking sessions with either a non-menthol control, menthol, or synthetic cooling agent cigarette condition once weekly (QW) over 3 weeks on study. Participants also participate in an ad libitum smoking session with either their usual brand cigarette or the study cigarette condition at the end of each study visit. Participants also undergo nasal swab collection over 5-10 minutes and spirometry and airwave oscillometry testing over 5-10 minutes pre- and post-smoking session at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 - 29 years
* Established cigarette user
* Willing to provide informed consent and abstain from using tobacco products 12 hours prior to the three lab sessions
* Read and speak English

Exclusion Criteria:

* Recently coronavirus disease 2019 positive (COVID-19+) or a recent COVID-19 hospitalization
* Self-reported unstable or significant psychiatric conditions
* History of cardiac event or distress within the past 3 months
* Are currently pregnant, planning to become pregnant, or breastfeeding
* Currently attempting to quit using combustible tobacco products
* Have suffered from any serious lung disease or infection in the past 30 days

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Cigarette Chemical Contents | Up to end of study, estimated 1 year
  Tobacco samples from all three study cigarette types (menthol, non-menthol, synthetic cooling agent) will be extracted with isopropanol containing carvacrol. Nicotine, menthol, WS-3, WS-5, WS-12, and WS-23 amounts (mass) present in the different cigarettes will be quantified using gas chromatography mass spectrometry.
Impact of Cooling Effects on Demand via the Forced Choice Task | Up to end of study intervention, up to 3 weeks
  At each study visit, after the participant has smoked the study cigarette, the participant must choose between smoking the study cigarette again, or smoking one of their own, usual brand cigarettes. Within each arm, the proportion of participants who opt to continue smoking the study cigarette will be reported. This will measure if demand for the study cigarettes is great enough to overcome the desire for the participant's own preferred cigarettes.
Abuse Liability via Puff Topography | Up to end of study intervention, up to 3 weeks
  Will be measured with a topography device that records frequency, duration, and flow rate of cigarette puffs. These measures are combined to inform overall cigarette puff behavior. Greater frequency, duration, and flow rate of cigarette puffs suggest greater abuse liability.
Cigarette Appeal | Up to end of study intervention, up to 3 weeks
  Participants will complete the Appeal and Sensory Quality questionnaire after smoking each study cigarette. This questionnaire will ask participants to rate each study cigarette for appeal characteristics such as liking, willingness to use again, flavor intensity, pleasantness of taste, etc. on a scale of 0 (not at all)-100(extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Alayna P Tackett, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu